CLINICAL TRIAL: NCT00936585
Title: NIH SUBSTUDY:Randomized, Double-blind, Placebo-controlled, Parallel-group Proof-of-concept Study to Assess the Efficacy, Safety and Tolerability of Two Single Infusions of AIN457 in Patients With Moderate to Severe Active Crohn's Disease
Brief Title: NIH Substudy of AIN457 (Anti-IL-17 Monoclonal Antibody) for Treatment of Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted by the sponsor
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 090175; 09-I-0175 (Other: NIAID)
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Colitis; Crohn's Disease; Inflammatory Bowel Disease
Keywords: Crohn's Disease; Infusion; Anti IL-17 Monoclonal Antibody; Placebo; Crohn Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis; Crohn Disease; Inflammatory Bowel Diseases | interventions — Monitoring, Immunologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunologic Monitoring (Other): Blood draws and colonoscopy performed on patients enrolled in both intervention arms of the main study
  Interventions: Other: Immunologic Monitoring

INTERVENTIONS:
Other: Immunologic Monitoring — blood draws and colonoscopy before and after receiving study drug

SUMMARY:
The objective of this NIH-specific substudy is immunologic monitoring of cytokine and immune cell responses in subjects undergoing treatment with AIN457 (human monoclonal anti-human interleukin-17A) for moderate to severe Crohn's disease. Recent data suggests that interleukin-17 (IL-17) is an important mediator of inflammation in certain animal models of Crohn's disease, and treatment aimed at blocking the IL-23-IL-17 axis can ameliorate the inflammatory changes. In addition, elevated expression of IL-l7 has been found in the gut tissue of patients with active Crohn's disease. This substudy will measure changes in cytokine production, relevant RNA expression, and immune cell populations (in the periphery and lamina propria) for correlation with clinical outcomes in order to explore the mechanisms of therapeutic response.

DETAILED DESCRIPTION:
Purpose:

* Crohn's disease is an inflammatory bowel disease with major symptoms such as diarrhea and abdominal pain when the disease is in an active stage.
* AIN457 is a protein developed by NOVARTIS that is used to stop the action of Interleukin-17 (IL-17), a protein made by the body that contributes to many different kinds of inflammatory diseases, including Crohn's disease. AIN457 is being developed for the potential treatment of various inflammatory diseases like rheumatoid arthritis and psoriasis, but has not been tested for suitability in people with Crohn's disease.

Objectives:

* The main objective of the NIH substudy is to obtain additional blood and gut biopsy tissue for monitoring biochemical changes in immune variables in response to study drug or placebo.
* The main objective of the main multicenter study (sponsored by NOVARTIS) is to determine whether AIN457 is safe and effective in the treatment of Crohn's disease, and if effective, how long the effect will remain.

Eligibility:

- Important eligibility criteria to consider for patients to be enrolled in the AIN457 trial include:

Inclusion criteria:

* Male or female; 18-75 years old
* Diagnosis of Crohn's disease for at least 3 months prior to screening
* Moderate to severe active Crohn's disease at baseline, defined as: CDAI greater than or equal to 220 and less than or equal to 450
* Active disease despite prior treatment with stable dose of corticosteroids for 2 weeks, or immunosuppressant for at least 3 months (e.g. methotrexate, azathioprine).

Exclusion criteria:

* Subjects with symptoms associated with active bowel stricturing disease and pre-stenotic dilation on radiography.
* Fistulizing disease if complicated by sepsis and/or untreated abscess.
* Subjects with multiple bowel surgeries and clinically important short bowel syndrome defined as an inability to maintain caloric intake.
* Prior therapy with rituximab.
* Receiving corticosteroids dose equivalent to a > 40mg dose of prednisone per day.
* Subjects demonstrating clinical improvement due to other Crohn's therapy.
* Subjects with active or history of clinically significant cardiac abnormalities.

Design:

* For the NIH substudy, additional blood will be drawn and a colonoscopy will be performed before the first infusion and after the second infusion.
* The multicenter study plans to enroll seventy-two (72) subjects with moderate to severe active Crohn's disease that is not controlled by corticosteroids, immunosuppressant (e.g. methotrexate or purine metabolites) or anti-inflammatory treatment (e.g. 5-ASA). At baseline visit, if the eligibility of the subject is confirmed, the subject will be randomized (2:1 ratio) to receive either AIN457 or placebo administered as a 2 hours intravenous infusion. A total of two infusions will be given on day 1 and day 22 respectively.
* After infusions there will be a follow-up period of up to 18 weeks.
* Once this study is completed, an extension study will be conducted that will offer access to AIN457. Patients who complete the current study may be eligible to enter the extension study and receive therapy with AIN457.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female; 18-75 years old
  2. All female subjects must have negative pregnancy test results at screening and baseline. Women of childbearing potential (WoCBP) must be using simultaneously double-barrier or two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc. Hormone replacement as either oral or implantable is acceptable as one form), from the time of screening and for the duration of the study, through study completion and for 4 months following study completion.

     Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

     Postmenopausal females must have had no regular menstrual bleeding for at least two (2) years prior to initial dosing. Menopause will be confirmed by a serum FSH level of > 40 IU/L at screening. Pregnancy test will be required only at screening.

     Female subjects who report surgical sterilization must have had the procedure at least six (6) months prior to initial dosing. Surgical sterilization procedures should be supported with clinical documentation made available to the sponsor and noted in the Relevant Medical History/Current Medical Conditions section of the CRF.

     If female subjects have male partners who have undergone vasectomy, the vasectomy must have occurred more than six (6) months prior to first dosing.
  3. Male subjects willing to use simultaneously two acceptable methods of contraception (e.g. spermicidal gel plus condom) for entire duration of the study, up to the study completion visit and at least for 6 months following the completion of the study.

     Periodic abstinence and withdrawal are not acceptable methods of contraception.
  4. Diagnosis of Crohn's disease for at least 3 months prior to screening
  5. Confirmation of Crohn's disease by endoscopic or imaging examination
  6. Moderate to severe active Crohn's disease at baseline, defined as:

     --CDAI greater than or equal to 220 and less than or equal to 450
  7. Patients with active disease despite prior treatment with corticosteroids for at least 2 weeks, or immunosuppressants for at least 3 months.

     * Patients who are being treated with azathioprine, 6-MP or MTX are eligible but must have been on a stable dose for at least 10 weeks prior to baseline.
     * Patients treated with corticosteroids are eligible but must have been on stable doses of prednisolone not exceeding 40 mg for two weeks prior to baseline.
     * Patients who are being treated with immunosuppressants other than those listed above, such as cyclosporine, tacrolimus and mycophenolate, are not eligible. These subjects will be required to stop immunosuppressants prior to baseline. These patients are eligible after observing a wash out period as specified in Exclusion criterion #7.
  8. Absence of clinically relevant abnormalities for screening laboratory test results
  9. Able to communicate well with the investigator, and to understand and comply with the requirements of the study.
  10. Understand and sign the written informed consent.

EXCLUSION CRITERIA:

Subjects meeting any of the following criteria will be excluded from entry into or continuation in the study, unless sponsor approval is obtained:

1. Body Mass Index is greater than 34.
2. Positive Purified Protein Derivative (PPD) tuberculin skin test of greater than or equal to 5 mm at screening or 6 months prior to screening. A positive PPD test will be defined using the [MMWR 2000 guidance], summarized as criteria for tuberculin positivity by risk group.

   * A PPD test should not be done in subjects who had a tuberculosis vaccination in the past. These subjects will be eligible to participate if, according to local guidelines, latent tuberculosis can be excluded.
   * For those study sites using QuantiFeron test a positive test at screening will exclude the subject from the participation in the study.
   * If the result for either PPD or QuantiFeron test is indeterminate, the subject will be excluded.
3. Subjects with symptoms associated with active bowel stricturing disease and pre-stenotic dilation on radiographs.
4. Fistulizing disease if complicated by sepsis and/or untreated abscess.
5. Subjects with multiple bowel surgeries and clinically important short bowel syndrome defined as an inability to maintain caloric intake.
6. a. Concomitant treatment with anti-TNF-alpha therapy (or other biological therapy) and systemic immunosuppressive agents such as cyclosporine, mycophenolate, pimecrolimus, or tacrolimus, except azathioprine, its metabolite 6-MP and MTX.

   The following washout period will be required for subjects to be eligible to participate in the trial.
   * Three (3) months washout prior to baseline for certolizumab
   * Two (2) months washout prior to baseline for adalimumab, etanercept and infliximab
   * One (1) month washout prior to baseline for cyclosporine, mycophenolate, pimecrolimus, tacrolimus, and any other systemic immunosuppressants not listed under exclusion criterion # 7b

     6b. Patients who are being treated with azathioprine, 6-MP or MTX are eligible but must have been on a stable dose for at least 10 weeks prior to baseline and throughout the whole study period.
7. Prior therapy with rituximab.
8. Receiving corticosteroid dose equivalent to a greater than 40mg dose of prednisone per day.
9. Subjects demonstrating clinical improvement due to other Crohn's therapy.
10. Current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, psychiatric, or other disease which would make the subject unsuitable for the trial.
11. Subjects with active or history of clinically significant cardiac abnormalities, for example:

    * Requiring drugs with QT-prolonging properties (e.g. antiarrhythmic drugs, such as amiodarone, sotalol, dofetilide, quinidine, procainamide, disopyramide).
    * QTc greater than 450msec long QT-syndrome (own or with a family history) or with a family history of sudden unexplained death.
    * Left branch bundle block (LBBB), or subjects who have been hospitalized for heart failure of cardiac etiology, in the previous 6 months, and subjects who have significant and persistent left-ventricular dysfunction (LVEF less than 40%).
    * History of in the preceding 3 months, significant and persistent arrhythmias such as ventricular fibrillation or tachycardia, or atrial fibrillation or flutter.
    * Symptomatic coronary artery disease.
    * Presence of severe cardiac disease (New York Heart Association Classification greater than or equal to III) and/or abnormal ECG, considered by the investigator to be unsafe for the study.
12. Liver disease or liver injury as indicated by abnormal liver function tests such as SGOT (AST), SGPT (ALT), gamma-GGT, alkaline phosphatase, or serum bilirubin. The Investigator should be guided by the following criteria:

    * Any single parameter may not exceed 2 times the upper limit of normal (ULN). A single parameter elevated up to and including 2 times the ULN should be re-checked once more as soon as possible, and in all cases, at least prior to enrollment/randomization, to rule out lab error.
    * If the total bilirubin concentration is increased above 2 times the ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin. In any case, serum bilirubin should not exceed the value of 1.6 mg/dL (27 micromol/L).

    Re-check results must be within normal limits (or returning to within normal limits) in order for subject to qualify.
13. Total WBC count which falls outside the range of 4500-13,000/microL, or platelets less than 100,000/microL at screening.
14. History of severe hypersensitivity to any biological agents (antibody or soluble receptor), including serious allergic reaction (hypotension, wheezing, urticaria), lupus-like syndrome or demyelinating disease.
15. Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing or longer if required by local regulation.
16. Administration of live vaccines within 6-month prior to dosing.
17. History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
18. A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
19. Significant illness within the two weeks prior to dosing or any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study.
20. Subjects with:

    * History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine greater than 1.3 mg/dL or blood urea nitrogen (BUN) greater than 30 mg/dL, or the presence of greater than +1 albumin on the urinary dipstick.
    * Presence of proteinuria, active sediments, casts or WBCs in urine.
    * Evidence of urinary obstruction or difficulty in voiding at screening.
    * History of renal trauma, glomerulonephritis, or subject with one kidney.
21. History of malignancy (other than basal cell carcinoma or adequately treated carcinoma-in-situ of the cervix).
22. Unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins.
23. Conditions associated with an immune-compromised condition such as recent surgical procedure; or history of drug or alcohol abuse within the 12 months prior to dosing. Subjects who are unable to discontinue analgesic medications containing opiates and opioids, as well as cannabinoids for medical use.
24. Participation in any clinical investigation within four (4) weeks prior to initial dosing or five half-lives of the investigational agent, whichever is longer, and for any other limitation of participation based on local regulations.

NIH EXCLUSION CRITERIA:

1. Platelet count less than 100,000 mm(3)
2. Prothrombin Time International Normalized ration (PT INR) greater than 1.3 or Partial Thromboplastin Time (PTT) 3 sec than control

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Yao, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abdul-Baki H, ElHajj I, El-Zahabi LM, Azar C, Aoun E, Zantout H, Nasreddine W, Ayyach B, Mourad FH, Soweid A, Barada KA, Sharara AI. Clinical epidemiology of inflammatory bowel disease in Lebanon. Inflamm Bowel Dis. 2007 Apr;13(4):475-80. doi: 10.1002/ibd.20022. PMID 17206720
- [Background] Baumgart DC, Sandborn WJ. Inflammatory bowel disease: clinical aspects and established and evolving therapies. Lancet. 2007 May 12;369(9573):1641-57. doi: 10.1016/S0140-6736(07)60751-X. PMID 17499606
- [Background] Best WR, Becktel JM, Singleton JW, Kern F Jr. Development of a Crohn's disease activity index. National Cooperative Crohn's Disease Study. Gastroenterology. 1976 Mar;70(3):439-44. PMID 1248701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited using advertisements and from patient database of Crohn's patients seen at the NIH CC.
Pre-assignment Details: All patients who were enrolled in the main study to receive study drug were eligible for the sub-study. There was no randomization.
Groups:
- Immunologic Monitoring: All patients who were enrolled in the main study participated in the NIH sub study and underwent a colonoscopy and blood draw for research specimens for immunologic monitoring before and after study drug administration
Period: Overall Study
Arm/Group | Immunologic Monitoring
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Immunologic Monitoring: Patients who received both placebo and drug infusions underwent a colonoscopy and blood draw for research specimens for immunological monitoring.
Arm/Group | Immunologic Monitoring
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (0.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Data
Description: Changes in immunological parameters in blood and lamina propria immune cells
Time Frame: Baseline, 6 weeks
Population: All patients in the study were enrolled; not enough patients were enrolled to get enough data to analyze - THERE IS NO DATA as the samples were not processed because not enough patients were enrolled to make any comparison.
Arm/Group | Immunologic Monitoring
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Colonoscopy: Patients who received both placebo and drug infusions underwent a colonoscopy and blood draw for research specimens for immunological monitoring.
Arm/Group | Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The NIH sub study ended earlier than anticipated as the Novartis main study was terminated for futility. As a result, not enough patients were enrolled to perform any analysis of data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes